CLINICAL TRIAL: NCT00929474
Title: BOOST: Benefit of Frequent Optimization After Cardiac Resynchronization Therapy Device Replacement
Brief Title: BOOST - Benefit of Frequent Optimization After Cardiac Resynchronization Therapy Device Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRD466
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- QuickOpt (Experimental)
  Interventions: Device: QuickOpt - SJM CRT (Group 1)
- Control (Active Comparator)
  Interventions: Device: Control - SJM CRT (Group 2)

INTERVENTIONS:
Device: QuickOpt - SJM CRT (Group 1) — The patient's device is programmed to sequential Bi-V pacing mode with paced/sensed AV and V-V delays optimized using QuickOpt. For Group 1 patients, optimization using QuickOpt is performed at enrollment, 3, 6, 9 and 12 month visits.
  Arms: QuickOpt
Device: Control - SJM CRT (Group 2) — The patient's device is programmed to either simultaneous or sequential Bi-V pacing mode as per physician's discretion. The paced/sensed AV and V-V delays could be programmed empirically or optimized using any non-intracardiac electrogram (IEGM) based method as per sites standard of care. However, the Group 2 patients can be optimized only once within the first 4 weeks post CRT replacement. Any paced/sensed AV and V-V delay optimizations performed after 4 weeks post CRT replacement in Group 2 patients will be considered a protocol deviation.
  Arms: Control

SUMMARY:
Cardiac resynchronization therapy (CRT) has shown improvement in mortality and morbidity in patients with left ventricular systolic dysfunction and congestive heart failure. Additionally in CRT patients it has been demonstrated that optimizing paced/sensed atrioventricular (AV) and interventricular (V-V) timings leads to immediate hemodynamic benefits and further improves cardiac function. Recent studies have shown that optimal paced/sensed AV and V-V delays change over time, which raises the question of how often optimization should be repeated. Thus, frequent re-optimization of these delays might be beneficial for maintaining significant improvement of cardiac function. However, it remains to be evaluated whether timing optimization may be beneficial on patients who have received CRT for a number of years and are now having the CRT device replaced.

DETAILED DESCRIPTION:
* This is a prospective, randomized, and multicenter study
* Patients who have received a replacement St. Jude Medical(SJM) CRT device, either CRT-P or CRT-D, within the last two weeks post CRT replacement will be considered for enrollment in the study.
* Baseline measurements will be performed at the time of enrollment.
* Patients are followed up to 12 months post CRT replacement with data collected at 3, 6, 9 and 12 months post CRT replacement.
* Patients will be randomized at enrollment to either Group 1 (use of SJM algorithm to optimize programming) or Group 2 ("Control").

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent a CRT replacement within the last two weeks, triggered by either the elective replacement indicator (ERI)/end of life (EOL), or by receiving a CRT-D device as an upgrade from a CRT-P device.
* Patient has received an FDA approved SJM CRT device as a replacement to the old CRT device within the last two weeks.
* Patient has the ability to complete a 6-minute hall walk without any assistance.
* Patient is willing to provide written informed consent.
* Patient has the ability to independently comprehend and complete a QOL questionnaire.
* Patient is geographically stable and is willing to comply with the required follow-up schedule.

Exclusion Criteria:

* Patient had paced/sensed AV and/or V-V delay optimization using QuickOpt before CRT replacement.
* Patient had any paced/sensed AV and/or V-V delay optimization within 3 months before CRT replacement.
* Patient has an ability to walk ≥ 450 meters (≥ 1476 feet) in 6 minutes.
* Adequate patient's echocardiography/Doppler images will not be available.
* Patient is expected to receive a heart transplant during the duration of the study.
* Patient has an epicardial ventricular lead system (Active or Inactive).
* Patient has limited intrinsic atrial activity (≤ 40 bpm).
* Patient has persistent or permanent atrial fibrillation (AF).
* Patient has 2° or 3° heart block.
* Patient's life expectancy is less than 1 year.
* Patient is less than 18 years old.
* Patient is pregnant.
* Patient is on IV inotropic agents 1 month prior to CRT replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Hattiesburg Clinic, P.A./Southern Heart Center, Hattiesburg, Mississippi

RESULTS

PARTICIPANT FLOW:
Groups:
- QuickOpt: QuickOpt - St. Jude Medical (SJM) cardiac resynchronization therapy (CRT) (Group 1) : The patient's device is programmed to sequential Bi-V pacing mode with paced/sensed atrio-ventricular (AV) and V-V delays optimized using QuickOpt. For Group 1 patients, optimization using QuickOpt is performed at enrollment, 3, 6, 9 and 12 month visits.
- Control: Control - SJM CRT (Group 2) : The patient's device is programmed to either simultaneous or sequential Bi-V pacing mode as per physician's discretion. The paced/sensed AV and V-V delays could be programmed empirically or optimized using any non-intracardiac electrogram (IEGM) based method as per sites standard of care. However, the Group 2 patients can be optimized only once within the first 4 weeks post CRT replacement. Any paced/sensed AV and V-V delay optimizations performed after 4 weeks post CRT replacement in Group 2 patients will be considered a protocol deviation.
Period: Overall Study
Arm/Group | QuickOpt | Control
Started | 8 | 9
Completed | 0 | 0
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QuickOpt | Control | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (10.2) | 77.7 (9.8) | 76 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Stroke Volume (SV) Measured by Aortic Velocity Time Integral (AoVTI)
Description: The BOOST study is prematurely terminated so there were no enough numbers of patients to have a meaningful measurement.
Time Frame: 12 months
Population: The BOOST study is prematurely terminated so there were no meaningful measurement from the study.
Arm/Group | QuickOpt | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | QuickOpt | Control
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QuickOpt (N=8) | Control (N=9)
Inappropriate therapy delivery (Cardiac disorders) | 0 (0) | 1 (1) — Implantable Cardioverter Defibrillator Therapy delivered of non-ventricular rhythm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No